CLINICAL TRIAL: NCT02962180
Title: Transplantation With Dermarolling System of Basal Cell Layer Suspension Obtained by Soft Trypsinisation in Vitiligo Lesion
Brief Title: Transplantation of Basal Cell Layer Suspension Using Derma-rolling System in Vitiligo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohammed V Souissi University (Other)
Responsible Party: Principal Investigator, BENZEKRI LAILA, PhD, Mohammed V Souissi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOHAMMED V UNIVERSITY
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Vitiligo
Keywords: derma-rolling system, vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Dermabrasion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm study (Experimental): Dermabrasion with dermaroller of basal cell layer suspension obtained by soft trypsinisation in vitiligo lesion.
  Interventions: Device: Dermabrasion with dermaroller

INTERVENTIONS:
Device: Dermabrasion with dermaroller — o The dermaroller is passed on the treated depigmented area. This technique is based on tiny microwounds performed using 540 microneedles (0.2mm length) which should allow the penetration of the suspension cells into the epidermis to obtain a good repigmentation.

SUMMARY:
Actually the methods for melanocyte delivery are invasive and often sophisticated. The dermarolling system with needles causing tiny microinjuries in the epidermis could offer a minimally invasive and painless method of melanocyte transplantation. The purpose of the study is to develop a new and simple method for transepidermally delivering keratinocytes and melanocytes into vitiligo skin.

DETAILED DESCRIPTION:
Condition: stable lesion of non segmental and segmental vitiligo of adults.

Background: The best method to transepidermally deliver isolated cells (melanocytes) is not yet defined. Microneedle treatment of the " ex vivo " human skin caused many thin vertical epidermodermal fissures and a variable depth of injury into the dermis regarding the length of the needles. This kind of treatment could be able to create small epidermal defects which allows to deliver melanocytes to an epidermal site. An approach to replenish melanocytes by injection of dissociated epidermal cell suspension with a syringe was recently successfully used. So, we hypothesize that the use of dermaroller with 0.2mm needle length which causes tiny microinjuries strictly in the epidermis could offer a simple, minimally invasive and painless method of melanocyte transplantation.

Main objective: To demonstrate the efficacy and the interest of dermaroller use with 0.2mm needle length in the transplantation of basal cell layer suspension in the epidermis of depigmented vitiligo skin.

Secondary objectives

1. To assess as control the effect of the use of dermaroller alone on the vitiligo lesion.
2. If transplantation is successful, to assess the duration needed to obtain a good coalescence and a complete repigmentation of the vitiligo lesion.

ELIGIBILITY:
Inclusion Criteria:

* Non segmental and segmental vitiligo lesions stable for a minimum of 1 year prior surgery
* Men and women aged over 18 years of age
* The lesion area must be 2cm2< lesion< 15cm2
* Absence of infected lesion

Exclusion Criteria:

* Actively spreading vitiligo (unstable disease)
* Patient with history of melanoma
* Infected lesions
* Positive Koebner Phenomenon
* History of hypertrophic scars or keloid formation
* Treatment with immunosuppressive or cytotoxic medication the past year
* Pregnant women and patients aged less 18 years
* Patients with concomitant photosensitizing treatment
* Positive serology of herpes, HIV, hepatitis B and C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-11 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rate of repigmentation lesions | At 6 months
  Image analysis

SECONDARY OUTCOMES:
Global satisfaction expressed by the patient | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: laila benzekri, Principal Investigator — Mohammed V University
Locations (1):
- Department of Dermatology, Ibn Sina University Hospital, Rabat, Morocco, Morocco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khodadadi L, Shafieyan S, Sotoudeh M, Dizaj AV, Shahverdi A, Aghdami N, Baharvand H. Intraepidermal injection of dissociated epidermal cell suspension improves vitiligo. Arch Dermatol Res. 2010 Oct;302(8):593-9. doi: 10.1007/s00403-010-1034-7. Epub 2010 Apr 4. PMID 20364383